CLINICAL TRIAL: NCT02475993
Title: SMART Mobile Application Technology Utilization in the Treatment of Sickle Cell Disease Post Day Hospital Discharge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00062922
Record Dates: First submitted 2015-06-17; First posted 2015-06-19 (Estimated); Last update posted 2019-10-18 (Actual); Status verified 2019-09

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMART app (Experimental): SMART, a mobile phone-based self-monitoring service to enhance outpatient treatment in chronic illness will be tested for its utility to help reduce acute care utilization rates for patients given SMART following acute care visits at the Sickle Cell Day Hospital. SMART will enable symptom monitoring with a particular emphasis on pain measures, co-symptoms, and related interventions aided by provider daily monitoring and support guided by patient report via SMART to provide a Sickle Cell Disease Information interchange (SCDi) service. Instead of using their current routine of triaging phone messages daily, assessing patients' need for intervention, providers will instead monitor patients' entries via SMART daily.
  Interventions: Other: SMART app
- Standard of care control group (No Intervention): The control group will get standard of care, including a printed plan for medications to be taken, phone number to call for questions or issues, and the return date for visit

INTERVENTIONS:
Other: SMART app — Subjects assigned to the intervention group will be given the pre-programmed SMART app on an iPad mini loaned to you for use during the study along with the medication plan as outlined in the discharge instructions and an appointment within 12 days. This will include SCD-related medications. Subjects will be asked to log entries each time they take their medications and will be reminded by SMART to take their medications based on their advised schedule. Follow up appointment time and date are also programmed into SMART, and reminders are given to the subject 3 days prior and on the day of appointment. Compliance will also be confirmed by pill count of all medications at the 30-day visit.
  Arms: SMART app

SUMMARY:
The purpose of this study is to test a web-aided, mobile-based PHR (Personal Health Reporting) service to enhance SCD outpatient treatment after discharge from an acute care setting, such as Duke University Medical Center's Day Hospital. SMART is a new mobile application created by SickleSoft to increase patient involvement in their treatment and improve patient to doctor communication. SMART is a self-monitoring and management service for SCD patients and their treatment doctors. This study will test whether or not use of the SMART mobile application will help develop the type of patient-doctor relationships that lead to better health outcomes and a decrease in readmission to an acute care facility.

DETAILED DESCRIPTION:
All patients seen for acute care of painful episodes in our Adult Sickle Cell Day Hospital will be screened for eligibility. Currently, there are >450 patients actively followed by staff in our adult Comprehensive Sickle Cell Center, with an average of 60-70 patient day hospital visits per month.

Intervention and control group. Patients enrolled will be alternately assigned to each group to ensure randomization and equal numbers of patients to each arm. All patients will be given a return appointment within 12 days of Day Hospital visit. The control group will get standard of care, including a printed plan for medications to be taken, phone number to call for questions or issues, and the return date for visit.

SMART Overview. SMART, a mobile phone-based self-monitoring service to enhance outpatient treatment in chronic illness will be tested for its utility to help reduce acute care utilization rates for patients given SMART following acute care visits at the Sickle Cell Day Hospital. SMART will enable symptom monitoring with a particular emphasis on pain measures, co-symptoms, and related interventions aided by provider daily monitoring and support guided by patient report via SMART to provide a Sickle Cell Disease Information interchange (SCDi) service. Instead of using their current routine of triaging phone messages daily, assessing patients' need for intervention, providers will instead monitor patients' entries via SMART daily. Our current clinicians, a nurse practitioner or medical doctor, will review data generated from patients' reports, as well as patient phone calls. Data entered daily by patients will be viewable by our clinicians. Rather than only listening to voice mails, a clinician from our provider team will view an electronic record and communicate with patients electronically by push notification, text messaging, secure email, or via the app. Our clinicians may also call patients by telephone, as they would do as necessary when responding to voice mails. .

ELIGIBILITY:
Inclusion Criteria:

* documented Hgb SS, SC, or HgbS-beta0 thalassemia
* age 18 years old or older
* seen during an acute care visit at the Duke Day Hospital

Exclusion Criteria:

* incapable of giving informed consent
* greater than 20 acute care visits within the past year
* patients on chronic RBC transfusions (scheduled transfusions)
* patients admitted to the hospital from the day hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-07; Primary Completion 2017-09-14 (Actual); Study Completion 2017-09-14 (Actual)

PRIMARY OUTCOMES:
percentage of acute care utilization | 30 days following discharge from the day hospital

SECONDARY OUTCOMES:
percentage adherence to hydroxyurea (HU) administration | 30 days following discharge from the day hospital
percentage adherence to post-acute care out-patient follow up visit | 30 days following discharge from the day hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States